CLINICAL TRIAL: NCT01887028
Title: A Single-blind, Randomized Study to Compare Impacts of Intraperitoneal Pressure (8mmHg Versus 12 mmHg) and CO2 Gas (Cool, Dry CO2 Gas Versus Warmed; Humidified Co2 Gas) on Surgical Peritoneal Environment During Laparoscopic Surgery
Brief Title: Impacts of Intraperitoneal Pressure and CO2 Gas on Surgical Peritoneal Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CHU-0158
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Laparoscopic Hysteretctomy With Promontofixation
Keywords: Carbon deoxide pneumoperitoneum; Intraperitoneal pressure; Peritoneum; Gene expression; Post-operative recovery; Laparoscopic Humidification System

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 12mmHg intraperitoneal pressure (cool, dry CO2 gas )(n=20) (Experimental)
  Interventions: Device: Fisher and Paykel Humidifier (MR860AEU)
- 12mmHg intraperitoneal pressure (warmed, humidified CO2 gas) (Other)
  Interventions: Device: Fisher and Paykel Humidifier (MR860AEU)
- 8mmHg intraperitoneal pressure with cool, dry CO2 gas (n=20) (Other)
  Interventions: Device: Fisher and Paykel Humidifier (MR860AEU)
- 8mmHg intraperitoneal pressure (warmed, humidified CO2 gas) (Other)
  Interventions: Device: Fisher and Paykel Humidifier (MR860AEU)

INTERVENTIONS:
Device: Fisher and Paykel Humidifier (MR860AEU) — Humidification to 98% relative humidity, and warming to 37 degrees C of laparoscopic insufflate. This will be done for the duration of the operation

SUMMARY:
Use lay language.

The primary purpose is to compare the impacts of intraperitoneal pressure (8mmHg versus 12 mmHg) and CO2 gas (cool, dry CO2 gas versus warmed, humidified CO2 gas) on gene expression in peritoneal tissues during laparoscopic surgery. We hypothesize that combined use of a low Intraperitoneal pressure (8mmHg) and warmed, humidified CO2 gas during CO2 pneumoperitoneum may be better in minimizing adverse effects on surgical peritoneal environment and improving clinical outcomes compared to the standard intraperitoneal pressure (12mmHg) and standard cool, dry CO2 gas.

DETAILED DESCRIPTION:
Patients undergoing laparoscopic hysterectomy with promontofixation are randomized into four groups: Group 1: 12mmHg intraperitoneal pressure with cool, dry CO2 gas (n=20), Group 2: 12mmHg intraperitoneal pressure with warmed, humidified CO2 gas (n=20), Group 3: 8mmHg intraperitoneal pressure with cool, dry CO2 gas (n=20), Group 4: 8mmHg intraperitoneal pressure with warmed, humidified CO2 gas (n=20).

Normal peritoneum is collected from the parietal wall at the beginning of laparoscopic surgery and at 1 and 2 hours. Expression of genes encoding components of the fibrinolytic system, extracellular matrix and adhesion molecules, and inflammatory cytokine signaling molecules in peritoneal tissues are measured by real-time PCR.

Quality of post-operative recovery by QoR-40, post-operative pain by Visual Analog Scale, per or post operative complications and intraoperative core temperature are assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years old
* Petients undergoing laparoscopic hysterectomy with promontofixation for uterine prolapse
* Menopaused
* ASA class I or II

Exclusion Criteria:

* Absolute contraindications to laparoscopy
* Previous history of pelvic surgery, endometriosis and/or infection
* Pathological peritoneal tissue
* BMI more than 30
* Height less than 150cm

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Expression of genes encoding components of the fibrinolytic system, extracellular matrix and adhesion molecules, and inflammatory cytokine signalling molecules in peritoneal tissues | at1 hour and 2 hours (day 1)

SECONDARY OUTCOMES:
Quality of post-operative recovery | at day 1
Post-operative pain | at day 1
Per or post operative complications | at day 1
Intraoperative core temperature | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Revaz BOTCHORISHVILI, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France